CLINICAL TRIAL: NCT03966183
Title: Early UVFP Management Based on Neurological Evidences (UVFP = Unilateral Vocal Fold Paralysis) (ION-UVFP) - Preliminary Study
Brief Title: Early UVFP Management Based on Neurological Evidences (ION-UVFP) - Preliminary Study
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/03OCT/365 - (1)
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Unilateral Vocal Cord Paralysis; Central Auditory Processing Disorder
MeSH Terms: conditions — Vocal Cord Paralysis; Language Development Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UVFP patients post thyroplasty: Patients in this group are adults who have undergone type I medialization thyroplasty (with Montgomery implant, silicone implant, follow-up of more than 3 months) as a definitive procedure following unilateral vocal fold paralysis.
- Control participants: The people in this group are control subjects of the same age, sex and manual laterality as the patients.

SUMMARY:
The purpose of this preliminary study is to help clarify our hypotheses for the longitudinal study by investigating the relationship between vocal cord paralysis and central auditory processes and thus the interpretation of auditory inputs into the central nervous system.

DETAILED DESCRIPTION:
A very recent study (Naunheim et al., 2018) shows that paralysis of a vocal cord can affect central auditory processes, which in turn would have a negative impact on motor control capabilities during voice production. This study was conducted in patients who had undergone Type I thyroplasty. To highlight these influences, the authors relied on behavioral tests of auditory perception and vocal production.

The investigators would like in this study, based on a similar and existing population at the Cliniques Universitaires Saint-Luc, to try to understand the changes observed clinically by proposing to perform vocal production tasks (also planned for the longitudinal study) in the MRI. The investigators would like to objectify the differences in the areas involved in the central auditory processes in comparison between patients and control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral paralysis in abduction of the vocal cords may be included in the study.
* Patients who undergone type I thyroplasty (with Montgomery implant) at least 3 months ago
* Control participants without voice disorder

Exclusion Criteria:

* Wear a pacemaker or other implanted devices (prostheses ...).
* Wear metal clips, metal in the head, or an adjustable brain drain.
* Wear non-removable dental appliances (except fillings).
* Wear cardiac valve prostheses.
* Have worked the metals.
* Have a tattoo containing metal particles.
* Have implanted jewelry (e.g., piercing).
* Being prone to epileptic seizures.
* Take medications that alter cortical excitability.
* Have had a brain surgery.
* Suffer from intracranial hypertension.
* Be pregnant or breastfeeding recently.
* Present allergies that are incompatible with the experimental protocol.
* Have an abnormal hearing loss in view of their age, identified with tonal and / or vocal audiometry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients who undergone type I thyroplasty (with Montgomery implant) at least 3 months ago after unilateral vocal fold paralysis
  * Control participants without voice disorder
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Voice quality | Min 3 months post thyroplasty
  Multidimensional voice assessment (Anamnestic interview, Maximum Phonation Time, Mean Air Flow, Mean subglottic pressure, Jitter, Shimmer, Noise-to-harmonic ratio, phonetogram, smoothed cepstral peak prominence, Voice Handicap Index - VHI-30, SF-36, EAT-10, GRBAS-I, Acoustic Voice Quality Index, Dysphonia Severity Index, Tonal and vocal audiometries)
Changes in the neuronal pathways involved in the processing of the auditory inputs | Max 6 months after involvement in the study
  Functional magnetic resonance imaging examination (tomodensitometry and connectivity)
Central auditory processes | Min 3 months post thyroplasty
  Auditory perception tasks performed using an audio headset (sound detection in noise, localization of a sound source, dichotic listening test, masking test, duration and frequency pattern test)

CONTACTS AND LOCATIONS:
Overall Officials: Gauthier Desuter, Principal Investigator — SSS/MEDE and SSS/IONS/NEUR
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No